CLINICAL TRIAL: NCT02016430
Title: Gut Flora Metabolite Reduction After Dietary Intervention (GRADY)
Acronym: GRADY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Wilson Tang, Staff Cellular and Molecular Medicine and Cardiovascular Medicine, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-863
Record Dates: First submitted 2013-12-15; First posted 2013-12-20 (Estimated); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Dietary Modification; Cardiovascular Risk Factor
Keywords: TMAO; Gut Flora; Dietary Intervention; Choline; Carnitine
MeSH Terms: interventions — trimethyloxamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MeLT Dietary intervention (Experimental): Mediterranean Low-TMAO (MeLT) diet. Used in cohorts 1, 2 and 3.
  Interventions: Behavioral: MeLT Dietary intervention
- TLC Dietary intervention (Experimental): Therapeutic Lifestyle Changes (TLC) diet. Used in cohorts 1, 2 and 3.
  Interventions: Behavioral: TLC Dietary intervention
- MeLT dietary intervention with TMAO (Experimental): Mediterranean Low TMAO diet with TMAO levels reported. Used in cohort 1 only.
  Interventions: Behavioral: MeLT dietary intervention with TMAO

INTERVENTIONS:
Behavioral: MeLT Dietary intervention — Mediterranean diet containing food with low TMAO content.
  Arms: MeLT Dietary intervention
Behavioral: TLC Dietary intervention — Standard American Heart Association (AHA) recommendations for dietary counseling.
  Arms: TLC Dietary intervention
Behavioral: MeLT dietary intervention with TMAO — Mediterranean diet containing food with low TMAO content with TMAO levels provided to the subject for guidance.
  Arms: MeLT dietary intervention with TMAO

SUMMARY:
Our group has recently identified the association between gut-flora-mediated carnitine and phosphatidylcholine metabolism, specifically trimethylamine-N-oxide (TMAO), and cardiovascular risk. This study investigates the ability for dietary intervention to modulate TMAO levels.

DETAILED DESCRIPTION:
This is a pilot human study to characterize the relationship between gut flora-associated TMAO generation and dietary intervention. The investigators hypothesize that tailored dietary interventions may help to reduce the ability for gut flora to generate TMAO in individuals with elevated TMAO levels. Specific aims include:

1. To investigate the proportion of subjects with persistently elevated circulating TMAO levels.
2. To compare the amount of TMAO generated from gut flora using stable-isotope-labelled choline, carnitine, and betaine in subjects with elevated versus normal circulating TMAO levels.
3. To evaluate the effect of dietary interventions on the amount of TMAO generated from gut flora using stable-isotope-labelled choline, carnitine, and betaine in subjects with elevated circulating TMAO levels.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1 Inclusion criteria:

* Men and women age 18 years or above.
* Elevated TMAO metabolizers (>5 µM) based on screening test and/or eGFR < 60 at most recent measurement.
* Willing to remain on aspirin or able to be off aspirin or aspirin products for 1 week prior to starting the study and staying on the same aspirin regimen during the duration of the study.
* Willing to sign the consent form and follow the study protocol, which includes a 12-week dietary modification.

Cohort 2 Inclusion criteria:

* Men and women age 18 years or above.
* Willing to remain on aspirin or able to be off aspirin or aspirin products for 1 week prior to starting the study and staying on the same aspirin regimen during the duration of the study.
* Willing to sign the consent form and follow the study protocol.
* eGFR values ranging from 16-59

Cohort 3 Inclusion criteria:

* Men and women age 18 years or above.
* Willing to remain on aspirin or able to be off aspirin or aspirin products for 1 week prior to starting the study and staying on the same aspirin regimen during the duration of the study.
* Willing to sign the consent form and follow the study protocol.

Exclusion Criteria (all cohorts):

* Significant chronic illness or end-organ dysfunction, including known history of uncompensated heart failure, renal failure, pulmonary disease, hematologic diseases.
* Active infection or received antibiotics within 2 months of study enrollment
* Use of over-the-counter probiotic within past month, or ingestion of yogurt within past 7 days
* Having undergone bariatric procedures or surgeries such as gastric banding or bypass.
* Pregnancy.
* Any condition which, in the judgment of the Investigator, would place a patient at undue risk by being enrolled in the trial, or cause inability to comply with the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2014-04-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in TMAO level | From baseline to 12 weeks follow-up
  The change in TMAO concentration measured in blood samples

CONTACTS AND LOCATIONS:
Overall Officials: W. H. Wilson Tang, MD, Principal Investigator — The Cleveland Clinic; Stanley L. Hazen, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Background] Wang Z, Klipfell E, Bennett BJ, Koeth R, Levison BS, Dugar B, Feldstein AE, Britt EB, Fu X, Chung YM, Wu Y, Schauer P, Smith JD, Allayee H, Tang WH, DiDonato JA, Lusis AJ, Hazen SL. Gut flora metabolism of phosphatidylcholine promotes cardiovascular disease. Nature. 2011 Apr 7;472(7341):57-63. doi: 10.1038/nature09922. PMID 21475195
- [Background] Koeth RA, Wang Z, Levison BS, Buffa JA, Org E, Sheehy BT, Britt EB, Fu X, Wu Y, Li L, Smith JD, DiDonato JA, Chen J, Li H, Wu GD, Lewis JD, Warrier M, Brown JM, Krauss RM, Tang WH, Bushman FD, Lusis AJ, Hazen SL. Intestinal microbiota metabolism of L-carnitine, a nutrient in red meat, promotes atherosclerosis. Nat Med. 2013 May;19(5):576-85. doi: 10.1038/nm.3145. Epub 2013 Apr 7. PMID 23563705
- [Background] Dalmeijer GW, Olthof MR, Verhoef P, Bots ML, van der Schouw YT. Prospective study on dietary intakes of folate, betaine, and choline and cardiovascular disease risk in women. Eur J Clin Nutr. 2008 Mar;62(3):386-94. doi: 10.1038/sj.ejcn.1602725. Epub 2007 Mar 21. PMID 17375117
- [Background] Bidulescu A, Chambless LE, Siega-Riz AM, Zeisel SH, Heiss G. Usual choline and betaine dietary intake and incident coronary heart disease: the Atherosclerosis Risk in Communities (ARIC) study. BMC Cardiovasc Disord. 2007 Jul 13;7:20. doi: 10.1186/1471-2261-7-20. PMID 17629908
- [Background] Tang WH, Wang Z, Levison BS, Koeth RA, Britt EB, Fu X, Wu Y, Hazen SL. Intestinal microbial metabolism of phosphatidylcholine and cardiovascular risk. N Engl J Med. 2013 Apr 25;368(17):1575-84. doi: 10.1056/NEJMoa1109400. PMID 23614584